CLINICAL TRIAL: NCT04831593
Title: The Rate of Full and Empty Stomach in a Large Cohort of Elective and Emergency Pediatric Patients by Preoperative Ultrasound Examination: a Prospective Observational Study
Brief Title: The Rate of Full and Empty Stomach in Elective and Emergency Pediatric Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ankara Children's Health and Diseases Hematology and Oncology Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Feyza Sever, Specialist physician, Ankara Children's Health and Diseases Hematology and Oncology Training and Research Hospital
Other Study IDs: 2019-167
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Ultrasound; Children; Surgery
Keywords: Ultrasound; Antrum; Children; Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Elective: In our clinic, pediatric patients who will undergo elective surgery, are performed gastric ultrasound before the operation. We aimed to see how often we met with empty and full stomach and to determine relationship between fasting time and qualitative assessment of gastric content in elective pediatric patients before general anesthesia.
  Interventions: Other: Group El
- Group Emergency: In our clinic, pediatric patients who will undergo emergency surgery, are performed gastric ultrasound before the operation. We aimed to see how often we met with empty and full stomach and to determine relationship between fasting time and qualitative assessment of gastric content in emergency pediatric patients before general anesthesia.
  Interventions: Other: Group Em

INTERVENTIONS:
Other: Group El — Gastric ultrasound is a point-of-care diagnostic tool to examine stomach contents and determine pulmonary aspiration risk at the bedside. Qualitative gastric sonography can determine the nature of gastric content ( empty, clear fluid or thick fluid/solid ) and quantitative gastric ultrasound can estimate the volume of gastric fluid.
  Other Names: Gastric ultrasound in elective pediatric patients before general anesthesia.
  Groups: Group Elective
Other: Group Em — Gastric ultrasound is a point-of-care diagnostic tool to examine stomach contents and determine pulmonary aspiration risk at the bedside. Qualitative gastric sonography can determine the nature of gastric content ( empty, clear fluid or thick fluid/solid ) and quantitative gastric ultrasound can estimate the volume of gastric fluid.
  Other Names: Gastric ultrasound in emergency pediatric patients before general anesthesia.
  Groups: Group Emergency

SUMMARY:
Background and Aim:

Pulmonary aspiration of gastric content in the perioperative period is rare, but it is an important cause of morbidity and mortality that anesthetists never want to encounter. Due to reasons such as emergency surgical procedures, communication problems with pediatric patients or their parents, impaired cognitive function, obesity, diabetes mellitus, chronic liver and kidney diseases, it is observed that there is sometimes inconsistency between the periods defined in the preoperative fasting guidelines in pediatric patients and the state of gastric content and volume encountered in clinical practice. There is a lack of data on children on this issue. In this study, primary we aimed to evaluate the incidence of empty and full stomach in pediatric patients who underwent elective and emergency surgery in our routine anesthesia practice. Also we want to determine the relationship between fasting time and qualitative assessment of gastric content. Secondary this study sought to examine whether correlation between gastric ultrasound finding and fasting time, and also to determine relationship with the current comorbidities.

Design:

This is a prospective, single blinded, observational study. The minimum sample size required to determine the prevalence of full stomach, 0.05, within the limits of ± 0.025 with 0.95 confidence, was calculated as 292.

When calculating with the proposed equation of n = 100 + 50i to determine the factors affecting by logistic regression (here i is the number of variables in the model), the minimum number of samples required for logistic regression analysis was calculated as 300 in case of 4 independent variables in the model. n=100+50*4= 300

Methods:

Pediatric patients younger than 18 yr old who are to undergo elective and emergency surgery under general anaesthesia at our hospital are enrolled in this prospective observational study between April and December 2021. Preoperative ultrasound examination of the gastric antrum are performed by one anesthesiologist who has been instructed and supervised by an experienced pediatric radiologist and who is blind to the patient's history. Ultrasonographic measurement of the gastric antral cross-sectional area (CSA) are performed in supine position and right lateral decubitus position (RLD). The gastric antrum is imaged in a sagittal plane, between the left lobe of the liver and the pancreas, at the level of the aorta, as previously described [1]. This examination allowed qualitative assessment of gastric contents according to the three-point grading scale previously described by Perlas and colleagues[2]. Grade 0 was defined by the absence of appearance of any content in a flat antrum in both the supine and the RLD positions. Grade 1 was defined by the appearance of any gastric content in the RLD position only, and Grade 2 was defined by the appearance of any content in both the RLD and the supine positions. The antral cross-sectional area is also calculated in both position, by measuring the longitudinal diameter (D1) and the anteroposterior diameter (D2) of the antrum, from serosa to serosa using this formula [3] Antral area= (π x D1 X D2) / 4. Patients' characteristic data ( age, gender, weight, height, BMI and ASA physical status classification), fasting duration, type of elective and emergency surgery, chronic disease and complications (regurgitation, pulmonary aspiration, etc.) that may develop during the peroperative period are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients younger than 18 yr old who are to undergo elective and emergency surgery under general anaesthesia are included in the study.

Exclusion Criteria:

* Exclusion criteria will be, having a nasogastric tube inserted and patient refusal.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric patients younger than 18 yr old who are to undergo elective and emergency surgery under general anaesthesia
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of full stomach | 30 minutes
  In our clinic, pediatric patients who will undergo emergency and elective surgery, are performed gastric ultrasound before the operation. We aimed to see how often we met with empty and full stomach in pediatric patients before general anesthesia.
The relationship between fasting time and qualitative assessment of gastric content | 30 minutes
  We would like to determine the relationship (and correlation with preoperative fasting guidelines) between the fasting time that pediatric patients and their parents reported to us and the qualitative assessment of gastric content in our clinical practice

SECONDARY OUTCOMES:
Demographic data and comorbidities | 30 minutes
  The secondary objective of this study is to examine correlation between gastric ultrasound finding and the demographic data ( age, gender, weight, height, BMI, ASA physical status classification), and type of elective and emergency surgery ) and current comorbidities of pediatric patients.

CONTACTS AND LOCATIONS:
Overall Officials: Feyza Sever, Principal Investigator — Ankara City Hospital Childrens' Hospital
Locations (1):
- Ankara City Hospital Childrens' Hospital, Ankara, Çankaya, Turkey (Türkiye)